CLINICAL TRIAL: NCT03245346
Title: Effects of Epidural Anesthesia and Analgesia on the Prognosis in Patients Undergoing Pancreatic Cancer Surgery: A Multi-center Randomized Controlled Trial
Brief Title: Effects of Epidural Anesthesia and Analgesia on the Prognosis in Patients Undergoing Pancreatic Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Changhong Miao, Director of Anesthesiology Department of Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FDUSCCA-1
Record Dates: First submitted 2017-08-02; First posted 2017-08-10 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Cancer of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Anesthesia, Epidural; Anesthesia, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEA+PCEA (Experimental): General anesthesia combined with epidural anesthesia will be performed during surgery and patient-controlled epidural analgesia (PCEA) will be provided after surgery.
  Interventions: Drug: GEA; Drug: PCEA
- GA+PCIA (Other): General anesthesia will be performed during surgery and patient-controlled intravenous analgesia (PCIA) will be provided after surgery.
  Interventions: Drug: GA; Drug: PCIA

INTERVENTIONS:
Drug: GEA — Thoracic epidural catheterization will be performed and epidural anesthesia will be maintained with 0.25% ropivacaine during surgery. General anesthesia will be maintained with inhalation (sevoflurane) and muscle relaxants will be administered when considered necessary.
  Other Names: General anesthesia combined with epidural anesthesia
  Arms: GEA+PCEA
Drug: PCEA — Patient-controlled epidural analgesia (0.15% ropivacaine infusion) will be provided after surgery.
  Other Names: Patient-controlled epidural analgesia
  Arms: GEA+PCEA
Drug: GA — General anesthesia will be maintained with inhalation (sevoflurane) and sufentanil infusion, and muscle relaxants will be administered when considered necessary.
  Other Names: General anesthesia
  Arms: GA+PCIA
Drug: PCIA — Patient-controlled intravenous analgesia (1ug/ml sufentanil) will be provided after surgery.
  Other Names: Patient-controlled intravenous analgesia
  Arms: GA+PCIA

SUMMARY:
The purpose of this randomized controlled trial is to investigate the effects of epidural anesthesia and analgesia on the overall survival，disease-free survival and recovery in patients undergoing pancreatic cancer surgery. This study will also evaluate the effects of this technique on neuroendocrine, stress and inflammatory response in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing elective pancreaticoduodenectomy for pancreatic cancer .
2. ASA statusⅠ-Ⅲ.
3. 18 years to 80 years （adults）.
4. Able to understand, communicate and sign an informed consent form.

Exclusion Criteria:

1. Laparoscopic surgery.
2. Preoperative chemotherapy or radiotherapy.
3. Pregnancy.
4. Allergic to any drugs used during the study.
5. Long-term receiving β-blockers.
6. Complicated with chronic inflammatory diseases, autoimmune diseases, or long-term receiving glucocorticoids or other immunosuppressants before surgery.
7. Abnormal coagulation functions (platelet count prior to surgery <100000/ μL , APTT value is more than the normal value, INR > 1.3 or clopidogrel that cannot be discontinued 7 days prior to surgery).
8. Complicated with severe heart disease (NYHA classification >3), severe renal insufficiency (serum creatinine >1.8mg/dL or receiving renal replacement therapy), severe hepatic disease (Child-Pugh classification

   = C), diabetes (fasting blood glucose not in the range of 3.9-13.8 mmol/L ), or acute infectious diseases (WBC>10000/μL) before surgery.
9. BMI > 35.
10. All contraindications to epidural anesthesia and analgesia.
11. Chronic opiate medication/drug abuse.
12. Complicated with severe mental illness, cognitive disorder or unable to collaborate during the study.
13. Refuse to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2021-12-18 (Estimated); Study Completion 2021-12-18 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | During 2 years after surgery
  Defined and calculated as the time from the date of surgery to death related to all reasons

SECONDARY OUTCOMES:
Disease-free survival (DFS ) | During 2 years after surgery
  Defined and calculated as the time from the date of surgery to the first time of pancreatic cancer recurrence or metastasis or cancer-related death
Postoperative pain score and side effects of patient-controlled analgesia | During the first 48 hours after surgery
  Assessed with visual analogue score ( 0 is no pain and 10 is the most severe pain)
Incidence of delirium | During the first 1 week after surgery
  Assessed for delirium using the 3D-CAM instrument
Incidence of persistent post-surgical pain (PPSP) after surgery | During 2 years after surgery
  Assessed with visual analogue score ( 0 is no pain and 10 is the most severe pain)
Length of stay in hospital after surgery and total costs after surgery | During the first 30 days after surgery
Return of bowel function | During the first 30 days after surgery
  Measured by the time of first flatus
Start of enteral tube feeding | During the first 30 days after surgery
  Measured by the time of first enteral tube feeding after surgery
Removal of Perianastomotic drains | During the first 30 days after surgery
Removal of Urinary drainage | During the first 30 days after surgery
Removal of nasogastric tube | During the first 30 days after surgery
Removal of enteral feeding tube | During the first 30 days after surgery
Blood level of neuroendocrine, stress and inflammatory response | During surgery and the first 24 hours after surgery (post-operative day 1)
  Changes of blood epinephrine, norepinephrine, cortisol, VEGF, interleukin-6 (IL-6)、interleukin-8 (IL-8), peripheral blood NLR ( neutrophil-lymphocyte ratio)
Serum CA19-9 、CA125、CEA、CA72-4、CA242、AFP、CA15-3、CA50 levels | During 2 years after surgery
Plasma levels of ropivacaine and sufentanil | During surgery and the first 24 hours after surgery (post-operative day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Changhong Miao, Principal Investigator — Fudan University; Qianjin Liu, Study Director — Washington University School of Medicine
Locations (3):
- China (3):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Fudan University Huashan Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Zhang H, Qu M, Guo K, Wang Y, Gu J, Wu H, Zhu X, Sun Z, Cata JP, Chen W, Miao C. Intraoperative lidocaine infusion in patients undergoing pancreatectomy for pancreatic cancer: a mechanistic, multicentre randomised clinical trial. Br J Anaesth. 2022 Aug;129(2):244-253. doi: 10.1016/j.bja.2022.03.031. Epub 2022 Jun 11. PMID 35697547